CLINICAL TRIAL: NCT01331200
Title: Early Mobilization of Ischemic Stroke Patients Within 24-hours After Intravenous-tPA Infusion.
Brief Title: Early Mobilization of Ischemic Stroke Patients Within 24-hours After Intravenous-Tissue Plasminogen Activator (IV-tPA)
Acronym: EMISTPA
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Scott Arnold, PT, Mayo Clinic Florida
Other Study IDs: 10-007822
Record Dates: First submitted 2011-02-04; First posted 2011-04-07 (Estimated); Last update posted 2013-02-27 (Estimated); Status verified 2013-02

CONDITIONS: Ischemic Stroke
Keywords: ischemic stroke; tissue plasminogen activator; early mobilization; patient safety; length of stay
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to study the safety and feasibility of mobilization of acute ischemic stroke patients treated with IV-tPA between 12-24 hours of treatment.

DETAILED DESCRIPTION:
Abstract:

Introduction

Historical precedence exists demonstrating that early intensive care unit (ICU) mobilization of patients reduces risks of complication and lengths of hospital stay, and may improve long-term health status of patients.

Objective

To determine the safety of early mobilization by physical and/or occupational therapy in acute ischemic stroke patients within 24-hours of IV-tPA infusion and to examine if early mobilization leads to shortened ICU and hospital length of stay.

Methods

Prospective study of incidence of adverse response and functional mobility status of study patients mobilized by occupational and/or physical therapy between 12- 24 hours after IV-tPA infusion with comparison of ICU and hospital Length of Stay data between study group and pre-study patients who were mobilized by occupational and/or physical therapy services at no pre-determined time after IV-tPA infusion. Additionally, patients will be contacted by study personnel approximately 3 to 5-days and 30-days post-infusion for completion of Modified Rankin Scale stroke disability survey as follow up of stroke recovery.

Setting

Medical and surgical intensive care units at Mayo Clinic Florida.

Patients

All patients with acute ischemic stroke who receive intravenous tissue plasminogen activator (IV-tPA) infusion, survive to discharge from the hospital, are hemodynamically stable, and are mobilized by physical and/or occupational therapy within 24 hours post-tPA infusion.

ELIGIBILITY:
Inclusion Criteria:

* Patients post acute ischemic stroke that have been treated with intravenous tissue plasminogen activator (IV-tPA)
* 13 hours have elapsed since initiation of intravenous TPA infusion
* Patients are hemodynamically stable (e.g., not on vasopressors or antihypertensive drips or requiring multiple IV PRN boluses of either medication)
* Patient is able to actively engage in the evaluation

Exclusion Criteria:

* Patients with femoral sheaths or recent removal of femoral sheaths
* Patients who are hemodynamically unstable, with active bleeding from lines, catheters, INT site or wounds or angioedema
* Electrocardiogram showing (HR>100)
* Vital signs (HR > 100, SBP <90 or >180, DBP <70 or > 105)
* Patients experiencing marked diaphoresis, facial pallor, intense anxious or painful facial expression (especially in aphasic patients)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients experiencing acute ischemic stroke who receive intravenous tissue plasminogen activator (IV-tPA) infusion, survive to discharge from the hospital, are hemodynamically stable, and are mobilized by physical and/or occupational therapy within 24 hours post-tPA infusion.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2011-01; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Level of Patient Disability post-TPA Infusion. | 30-days post-IV tPA infusion
  Study participants will be contacted at approximately 3 to 5-days and 30-days post-IV tPA infusion to capture level of disability by use of Modified Rankin Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Scott M Arnold, PT, Principal Investigator — Mayo Clinic; Olivia S Chavez, MS, OTR/L, Principal Investigator — Mayo Clinic; William D Freeman, MD, Principal Investigator — Mayo Clinic; James Meschia, MD, Principal Investigator — Mayo Clinic; Lesia Mooney, RN, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Hospital, Jacksonville, Florida, United States